CLINICAL TRIAL: NCT06951945
Title: Multiple Dose Study to Investigate the Safety, Tolerability, Pharmacokinetics, and Efficacy of THDBH120 in Chinese Patients With Obesity: A Randomized, Bouble-Blind, Placebo-Controlled Phase Ib Trial
Brief Title: Multiple Dose Study to Investigate the Safety, Tolerability, Pharmacokinetics, and Efficacy of THDBH120 in Chinese Patients With Obesity
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Tonghua Dongbao Pharmaceutical Co.,Ltd (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: THDBH120L107
Record Dates: First submitted 2025-04-23; First posted 2025-04-30 (Actual); Last update posted 2025-04-30 (Actual); Status verified 2025-04

CONDITIONS: Obesity
MeSH Terms: conditions — Obesity

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- THDBH120 injection (Experimental)
  Interventions: Drug: THDBH120 injection
- Placebo of THDBH120 injection (Placebo Comparator)
  Interventions: Drug: Placebo of THDBH120 injection

INTERVENTIONS:
Drug: THDBH120 injection — Participants received THDBH120 by subcutaneous injection.
  Arms: THDBH120 injection
Drug: Placebo of THDBH120 injection — Participants received placebo by subcutaneous injection.
  Arms: Placebo of THDBH120 injection

SUMMARY:
The aim of this trial is to investigate the safety, tolerability, pharmacokinetics, and efficacy of THDBH120 injection in participants with obesity. This study includes three multiple-ascending dose cohorts.

ELIGIBILITY:
Inclusion Criteria:

* Age between 18 and 65 years (inclusive), male or female;
* Body mass index (BMI) ≥ 28 kg/m²;
* Diet and exercise control for at least 3 months before screening visit, and less than 5% self-reported change within the last 3 months.

Exclusion Criteria:

* Type 1 diabetes, type 2 diabetes, gestational diabetes, or other types of diabetes;
* History of obesity attributable to endocrine diseases, monogenic mutations, or drug-induced causes, such as hypothalamic obesity, pituitary obesity, hypothyroid obesity, Cushing's syndrome, insulinoma, acromegaly, or hypogonadism; or weight gain resulting from increased non-fat mass (e.g., edema);
* Presence of uncontrolled hypertension at screening: systolic blood pressure ≥160 mmHg and/or diastolic blood pressure ≥100 mmHg;
* Prolonged QTcF interval on 12-lead ECG at screening (QTcF≥450 ms for males, >470 ms for females), PR interval >200 ms, or the presence of long QT syndrome, second- or third-degree atrioventricular block, left or right bundle branch block, Wolff-Parkinson-White syndrome, or any other clinically significant arrhythmias (except sinus arrhythmia).

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 36 (Actual)
Dates: Start 2024-07-18 (Actual); Primary Completion 2024-12-23 (Actual); Study Completion 2024-12-23 (Actual)

PRIMARY OUTCOMES:
Number of Participants with One or More Adverse Event(s) and Serious Adverse Event(s) | 78 days

SECONDARY OUTCOMES:
Pharmacokinetics (PK): Area Under the Concentration Versus Time Curve (AUC) of THDBH120. | Day 1 Pre-dose through Day 43
Pharmacokinetics (PK): Maximum Drug Concentration (Cmax) of THDBH120 | Day 1 Pre-dose through Day 43
Change From Baseline in Body Weight | 43 days
Number of Participants With Anti-THBHD120 Antibodies | 78 days

CONTACTS AND LOCATIONS:
Locations (2):
- China (2):
  - The First Affiliated Hospital of Bengbu Medical University, Anhui
  - Hangzhou First People's Hospital, Zhejiang

IPD SHARING:
Plan to Share IPD: No